CLINICAL TRIAL: NCT05272150
Title: A Phase 3b, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety and Efficacy of Guselkumab for the Treatment of Participants With Skin of Color Who Have Moderate-to-Severe Plaque Psoriasis and/or Moderate-to-Severe Scalp Psoriasis
Brief Title: Study of Guselkumab in Skin of Color Participants With Moderate-to-severe Plaque and/or Scalp Psoriasis
Acronym: VISIBLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109163; CNTO1959PSO3018 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-03-01; First posted 2022-03-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Plaque Psoriasis; Scalp Psoriasis
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Moderate-to-severe Plaque Psoriasis (Experimental): Participants will receive either guselkumab subcutaneously (SC) or placebo SC. Placebo participants will then crossover to receive guselkumab SC.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Cohort B: Moderate-to-severe Scalp Psoriasis (Experimental): Participants will receive either guselkumab SC or placebo SC. Placebo participants will then crossover to receive guselkumab SC.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Participants will receive guselkumab as subcutaneous injection.
  Other Names: CNTO1959; Tremfya
Drug: Placebo — Participants will receive placebo as subcutaneous injection.

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab treatment versus placebo in skin of color participants with predominant moderate-to-severe body psoriasis or predominant moderate-to-severe scalp psoriasis by assessing improvements in the signs and symptoms of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque psoriasis (with or without psoriatic arthritis [PsA]) for at least 6 months before the first administration of study drug
* Self-identify as non-white or non-caucasian
* Be a candidate for phototherapy or systemic treatment for psoriasis
* Have an involved body surface area (BSA) greater than or equal to (>=) 10 percent (%), psoriasis area and severity index (PASI) >=12, investigator global assessment (IGA) >=3 at screening and at baseline (Cohort A), or have a scalp surface area >=30%, psoriasis scalp severity index (PSSI) >=12, scalp specific investigator global assessment (ss-IGA) >=3, and one plaque outside of the scalp at screening and at baseline (Cohort B)
* Agree not to receive a live virus or live bacterial vaccination during the study, or within 12 weeks after the last administration of study intervention
* Agree not to receive a Bacillus Calmette-Guérin (BCG) vaccination during the study, and within 12 weeks after the last administration of study intervention

Exclusion Criteria:

* Has a nonplaque form of psoriasis (example: erythrodermic, guttate, or pustular)
* Has received ustekinumab, ixekizumab, secukinumab, or brodalumab within 12 weeks of first dose of study drug
* Has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Participant has known allergies, hypersensitivity, or intolerance to guselkumab or its excipients
* Has or has had a serious infection (example: sepsis, pneumonia or pyelonephritis), or has been hospitalized or received intravenous antibiotics for an infection during the 2 months before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Cohort A: Percentage of Participants who Achieve Psoriasis Area and Severity Index (PASI) 90 Response at Week 16 | Week 16
  A PASI 90 response is defined as greater than or equal to (>=) 90 percent (%) improvement in PASI score from baseline. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Cohort A: Percentage of Participants who Achieve an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 16 | Week 16
  Percentage of participants with IGA score of 0 (cleared) or 1 (minimal) will be reported. The IGA documents the investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Cohort B: Percentage of Participants who Achieve Psoriasis Scalp Severity Index (PSSI) 90 Response at Week 16 | Week 16
  A PSSI 90 response is defined as >=90% reduction in PSSI score from baseline. The PSSI measures the extent of psoriasis involvement and the severity of erythema, infiltration, and desquamation of the scalp. Involved scalp area is measured on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved), clinical symptoms are each rated from 0 (absent) to 4 (severest possible). Involvement and severity of psoriasis for the PSSI is scored by physicians using a scale from 0 to 72, where 0=no psoriasis, and higher scores indicating more severe disease.
Cohort B: Percentage of Participants who Achieve Scalp-specific Investigator Global Assessment (ss-IGA) Score of Absence of Disease (0) or Very Mild Disease (1) at Week 16 | Week 16
  Percentage of participants with ss-IGA score 0 (absence of disease) or 1 (very mild disease) will be reported. The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: absence of disease (0), very mild disease (1), mild disease (2), moderate disease (3), and severe disease (4).

SECONDARY OUTCOMES:
Cohort A: Percentage of Participants who Achieve IGA Score of Cleared (0) at Week 16 | Week 16
  Percentage of participants with IGA score 0 (cleared) will be reported. The IGA documents the investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Cohort A: Percentage of Participants who Achieve PASI 100 Response at Week 16 | Week 16
  A PASI 100 response is defined as 100% improvement in PASI score from baseline. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Cohort A: Change from Baseline in PASI Score at Week 16 | Baseline and Week 16
  Change from baseline in PASI score at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the total PASI score. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Cohort A: Change from Baseline in Body Surface Area (BSA) at Week 16 | Baseline and Week 16
  Change from baseline in BSA at Week 16 will be reported. The BSA is a measurement of involved skin over the whole body. The overall BSA affected by psoriasis is estimated based on the participant's handprint (defined as the entire palmar surface of the hand including fingers).
Cohort A: Time to >=90% Reduction in PASI Score | Up to Week 16
  Time to >=90% reduction in PASI score will be reported which is defined as time to achieve >=90% improvement in PASI. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Cohorts A and B: Change from Baseline in Dermatology Life Quality Index (DLQI) Score at Week 16 | Baseline and Week 16
  Change from baseline in DLQI score at Week 16 will be reported. The DLQI is a dermatology specific quality of life instrument designed to assess the impact of dermatologic disease on a participant's quality of life (QoL). It is a 10 item patient-reported outcome(s) (PRO) questionnaire that, in addition to evaluating overall QoL, can be used to assess 6 different aspects that may affect QoL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The DLQI produces a numeric score that can range from 0 to 30. A higher score indicates more severe disease.
Cohort A: Percentage of Participants who Achieve >= 4-point Reduction (Improvement) from Baseline in the Psoriasis Symptom and Sign Diary (PSSD) Itch Score at Week 16, Among Participants with Baseline PSSD Itch >= 4 at Baseline | Week 16
  Percentage of participants who achieve >=4-point reduction (improvement) from baseline in PSSD itch score at Week 16 among participants with baseline PSSD itch >=4 at baseline will be reported. The PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefits. The participants are asked to answer the questions thinking about either the last 24 hours (24-hour recall version) or the last 7 days (7 days recall version). Both versions include 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Two subscores will be derived, each ranging from 0-100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Cohorts A and B: Percentage of Participants who Achieve a PSSD Symptom Score of 0 at Week 16, Among Randomized Participants with Baseline PSSD Symptom Score >=1 | Week 16
  Percentage of participants who achieve a PSSD symptom score of 0 at Week 16 among randomized participants with baseline PSSD symptom score >=1 will be reported. The PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefits. The participants are asked to answer the questions thinking about either the last 24 hours (24-hour recall version) or the last 7 days (7 days recall version). Both versions include 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Two subscores will be derived, each ranging from 0-100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Cohorts A and B: Change from Baseline in PSSD Symptom Score at Week 16 | Baseline and Week 16
  Change from baseline in PSSD symptom score at Week 16 will be reported. The PSSD includes PRO questionnaires designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefits. The participants are asked to answer the questions thinking about either the last 24 hours (24-hour recall version) or the last 7 days (7 days recall version). Both versions include 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Two subscores will be derived, each ranging from 0-100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Cohort B: Percentage of Participants who Achieve ss-IGA Score of Absence of Disease (0) at Week 16 | Week 16
  Percentage of participants with ss-IGA score 0 (absence of disease) will be reported. The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: absence of disease (0), very mild disease (1), mild disease (2), moderate disease (3), and severe disease (4).
Cohort B: Change from Baseline in Scalp Surface Area (SSA) at Week 16 | Baseline and Week 16
  Change from baseline in SSA at Week 16 will be reported. The SSA is a measurement of involved skin on the scalp. The overall SSA affected by psoriasis will be estimated based on the participant's thumb.
Cohort B: Percentage of Participants who Achieve PSSI 100 Response at Week 16 | Week 16
  A PSSI 100 response is defined as 100% reduction in PSSI score from baseline. The PSSI measures the extent of psoriasis involvement and the severity of erythema, infiltration, and desquamation of the scalp. Involved scalp area is measured on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved), clinical symptoms are each rated from 0 (absent) to 4 (severest possible). Involvement and severity of psoriasis for the PSSI is scored by physicians using a scale from 0 to 72, where 0=no psoriasis, and higher scores indicating more severe disease.
Cohort B: Change from Baseline in PSSI Score at Week 16 | Baseline and Week 16
  Change from baseline in PSSI score at Week 16 will be reported. The PSSI measures the extent of psoriasis involvement and the severity of erythema, infiltration, and desquamation of the scalp. Involved scalp area is measured on a scale from 0 (0% of scalp involved) to 6 (90-100% of scalp involved), clinical symptoms are each rated from 0 (absent) to 4 (severest possible).The PSSI total score is a composite score derived from the sum of the scores for erythema, induration and desquamation multiplied by the score for the extent of scalp area involved (percent of scalp involved). Involvement and severity of psoriasis for the PSSI is scored by physicians using a scale from 0 to 72, where 0=no psoriasis, and higher scores indicating more severe disease.
Cohort B: Time to >=90% Reduction in PSSI Score | Up to Week 16
  Time to >=90% reduction in PSSI score will be reported which is defined as time to achieve >=90% improvement in PSSI. The PSSI measures the extent of psoriasis involvement and the severity of erythema, infiltration, and desquamation of the scalp. Involvement and severity of psoriasis for the PSSI is scored by physicians using a scale from 0 to 72, where 0=no psoriasis, and higher scores indicating more severe disease.
Cohort B: Percentage of Participants with >= 4 Point Reduction (Improvement) from Baseline in the Scalp Itch NRS Score at Week 16, Among Participants with Baseline Scalp Itch >=4 at Baseline | Week 16
  Percentage of participants with >=4 point reduction (improvement) from baseline in scalp itch NRS score, among participants with scalp itch >=4 at baseline will be reported. The scalp itch NRS is a single-item scale that asks participants to rate the severity of their scalp itching due to psoriasis by considering their worst level of itching over the past 24 hours. The participants will be asked to assess scalp itch and select a number on a scale of 0-10, where "0" represents no scalp itch, and "10" represents the worst imaginable scalp itch.
Cohorts A and B: Number of Participants with Adverse Events (AEs) | Up to Week 116
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Cohorts A and B: Number of Participants with Serious Adverse Events (SAEs) | Up to Week 116
  SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (94):
- United States (79):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Cahaba Research Inc, Birmingham, Alabama
  - Stoll Dermatology, Beverly Hills, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Community Regional Medical Center, Fresno, California
  - Paul Wallace MD, Ladera Heights, California
  - The Grimes Center for Medical and Aesthetic Dermatology, Los Angeles, California
  - Care Access Research, Newport Beach, California
  - MedDerm Associates, San Diego, California
  - Synergy Clinical Research, San Francisco, California
  - Southern California Dermatology, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Center for Dermatology and Dermatologic Surgery, Washington D.C., District of Columbia
  - Skin Care Research, Boca Raton, Florida
  - Driven Research LLC, Coral Gables, Florida
  - Florida Academic Dermatology Centers, Coral Gables, Florida
  - Hollywood Dermatology and Cosmetic Surgery, Hollywood, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Tory P Sullivan M D PA, North Miami Beach, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Riverchase Dermatology and Cosmetic Surgery, Pembroke Pines, Florida
  - GCP Research, St. Petersburg, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Hamilton Dermatology Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Advanced Medical Research, Atlanta, Georgia
  - Skin Care Physicians of Georgia, Macon, Georgia
  - University Dermatology and Vein Clinic, Darien, Illinois
  - Northshore University Healthsystem, Skokie, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - Ds Research, Louisville, Kentucky
  - Callender Center for Clinical Research, Glenn Dale, Maryland
  - Care Access Research, Marriottsville, Maryland
  - DermAssociates, PC, Rockville, Maryland
  - Lawrence J Green MD LLC, Rockville, Maryland
  - Allcutis Research, Beverly, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - David Fivenson MD, Dermatology, Ann Arbor, Michigan
  - St Joseph Dermatology and Vein Clinic, Saint Joseph, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Henry Ford Medical Center, West Bloomfield, Michigan
  - Twin Cities Dermatology Center, Minneapolis, Minnesota
  - Skin Specialists, Omaha, Nebraska
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Hudson Dermatology & Skin Cancer Center, Hoboken, New Jersey
  - Schweiger Dermatology Group, Verona, New Jersey
  - Forest Hills Dermatology Group PLLC, Forest Hills, New York
  - MDCS Dermatology, New York, New York
  - Sadick Research Group, New York, New York
  - Markowitz Medical OptiSkin, New York, New York
  - Accellacare Research of Cary, Cary, North Carolina
  - Darst Dermatology, Charlotte, North Carolina
  - Dermatology Specialists, Charlotte, North Carolina
  - Accellacare of Raleigh, Raleigh, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - Advanced Dermatology and Skin Cancer Center, Boardman, Ohio
  - Wright State Physicians Health Center, Dayton, Ohio
  - Apex Dermatology Mayfield Heights, Mayfield Heights, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Schweiger Dermatology Group, Exton, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Dermatology and Laser Center of Charleston, Charleston, South Carolina
  - Palmetto Clinical Trial Services, LLC, Fountain Inn, South Carolina
  - Arlington Center for Dermatology, Arlington, Texas
  - Dermatology Treatment & Research Center, PA, Dallas, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce and Associates - The Center for Skin Research, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
- Canada (15):
  - Dermatology Research Institute Inc, Calgary, Alberta
  - Beacon Dermatology, Calgary, Alberta
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - Dr. Chih ho Hong Medical, Surrey, British Columbia
  - Dr. Lorne E. Albrecht, Surrey, British Columbia
  - CCA Medical Research Corporation, Ajax, Ontario
  - Dr Dusan Sajic Medicine Professional Corporation, Guelph, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North York Research Inc, North York, Ontario
  - JRB Research Inc, Ottawa, Ontario
  - Nectar Research Group Inc, Richmond Hill, Ontario
  - Canadian Dermatology Center, Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - FACET Dermatology, Toronto, Ontario
  - Research Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Alexis A, McMichael A, Soung J, Choi O, Alkousakis T, Alonso-Llamazares J, Shahriari M, Rodriguez AO, Bhutani T, Chan D, Rowland K, Sauder M, Hong HC, Yadav G, Yeung J, Jeyarajah J, Ma T, Gao LL, Park-Wyllie L, Green L, Lee M, Vashi N, Kindred C, Grimes P, Taylor SC, Desai SR; VISIBLE Trial Investigators. Guselkumab for Moderate to Severe Psoriasis Across All Skin Tones: Cohort A of the VISIBLE Randomized Clinical Trial. JAMA Dermatol. 2025 Sep 1;161(9):901-911. doi: 10.1001/jamadermatol.2025.1836. PMID 40560559
- [Derived] McMichael A, Shahriari M, Stein Gold L, Alkousakis T, Choi O, Bhutani T, Rodriguez AO, Tyring SK, Chan D, Rowland K, Albrecht L, Lynde C, Yadav G, Yeung J, Park-Wyllie L, Ma T, Jeyarajah J, Gao LL, Smith S, Moore AY, Vashi N, Kindred C, Grimes P, Desai SR, Taylor SC, Alexis A; VISIBLE Trial Investigators. Guselkumab for Moderate to Severe Scalp Psoriasis Across All Skin Tones: Cohort B of the VISIBLE Randomized Clinical Trial. JAMA Dermatol. 2025 Sep 1;161(9):912-922. doi: 10.1001/jamadermatol.2025.1849. PMID 40560554
- [Derived] Alexis A, McMichael A, Vashi N, Bhutani T, Rodriguez AO, Yeung J, Choi O, Chan D, Alkousakis T, Bronner DN, Park-Wyllie L, Gao LL, Grimes P, Shahriari M, Yadav G, Kindred C, Taylor SC, Desai SR. Improving Diversity in a Novel Psoriasis Study: VISIBLE as a Framework for Clinical Trial Quality Improvement. JAMA Dermatol. 2025 Mar 1;161(3):256-264. doi: 10.1001/jamadermatol.2024.5103. PMID 39661358